CLINICAL TRIAL: NCT02208700
Title: Efficacy of the Use of Enteral Feeding High in EPA,GLA and Antioxidants in LTAC Patients on Chronic Ventilation- a Pilot Study
Brief Title: Efficacy of Oxepa Enteral Feeding in LTAC (Long Term Acute Care Hospital) Patients on Chronic Ventilation- a Pilot Study
Acronym: ANUS1305
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grace Hospital, Cleveland, Ohio (Other)
Collaborators: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1141459
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Acute Lung Injury; Mechanical Ventilation Complication; Dietary Modification
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxepa (Experimental): Other: Therapeutic nutrition with EPA, GLA and antioxidants.
  Interventions: Other: Oxepa
- Jevity 1.5 (Active Comparator): Other: Jevity 1.5 Complete Balanced Nutrition with Fiber .
  Interventions: Other: Jevity 1.5

INTERVENTIONS:
Other: Oxepa — Therapeutic nutrition with EPA, GLA< and antioxidants
  Arms: Oxepa
Other: Jevity 1.5 — Complete balanced nutrition with a unique fiber blend
  Arms: Jevity 1.5

SUMMARY:
Patients with mechanical ventilation have shown improved weaning rates when enteral tube feeding high in EPA, GLA and antioxidants were fed to patients in the critical care setting.

LTAC Patients on chronic mechanical ventilation will have decreased days an mechanical ventilation, decreased mortality rates and decreased organ failure when fed an enteral product high in EPA, GLA and antioxidants compared to an isotonic high fiber enteral nutrition product.

ELIGIBILITY:
Inclusion Criteria:

>18 years old with Respiratory failure on mechanical ventilation with failure to wean Diagnosis of ARDS (Acute respiratory Distress Syndrome) Bilateral infiltrates -

Exclusion Criteria:

History Of pulmonary fibrosis, Terminal illness/ malignancies, <28 day life expectancy, Hemodialysis, Active bleeding or bleeding disorder: DIC ( Disseminated intravascular Coagulation), Sickle Cell Anemia, Hemophilia Hemorrhagic or ischemic stroke, Liver failure, Head trauma with Glasgow coma scale score of <5, Immunosuppression: WBC(White Blood Cell Count) <5000, HIV positive, use of immunosuppressant drugs, Pregnancy, and Heart Failure with EF(Ejection Fraction) <35%

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Length of days on mechanical ventilation | 14 days from start of enteral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Basma Ricaurte, MD, Principal Investigator — Grace Hospital
Locations (1):
- Grace Hospital, Cleveland, Ohio, United States